CLINICAL TRIAL: NCT05120336
Title: The Effects of Transcutaneous Vagus Nerve Stimulation on Motivation in Major Depressive Disorder
Brief Title: tVNS Effects on Motivation in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NBK_TUE004
Record Dates: First submitted 2021-10-18; First posted 2021-11-15 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder
Keywords: vagus nerve stimulation; food reward; anhedonia; vigor; reward learning; mood
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-depressed control participants: sham first, active taVNS second (Experimental): Non-depressed control participants receive sham stimulation in the first session (biphasic stimulation with a frequenyc of 25 Hz, 30s OFF/30s ON at the earlobe (sham) for 1.5 h). In a second identical session, they receive active stimulation with the same parameters (at the cymba conchae).
  Interventions: Device: transcutaneous vagus nerve stimulation; Device: sham stimulation
- Patients with major depressive disorders: sham first, active taVNS second (Experimental): participants with depression receive sham stimulation in the first session (biphasic stimulation with a frequenyc of 25 Hz, 30s OFF/30s ON at the earlobe (sham) for 1.5 h). In a second identical session, they receive active stimulation with the same parameters (at the cymba conchae).
  Interventions: Device: transcutaneous vagus nerve stimulation; Device: sham stimulation
- Patients with major depressive disorders: active taVNS first, sham second (Experimental): participants with depression receive active stimulation in the first session (biphasic stimulation with a frequenyc of 25 Hz, 30s OFF/30s ON at the cymba conchae (active) for 1.5 h). In a second identical session, they receive sham stimulation with the same parameters (at the earlobe).
  Interventions: Device: transcutaneous vagus nerve stimulation; Device: sham stimulation
- Non-depressed control participants: active taVNS first, sham second (Experimental): Non-depressed control participants receive active stimulation in the first session (biphasic stimulation with a frequenyc of 25 Hz, 30s OFF/30s ON at the cymba conchae (active) for 1.5 h). In a second identical session, they receive sham stimulation with the same parameters (at the earlobe).
  Interventions: Device: transcutaneous vagus nerve stimulation; Device: sham stimulation

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — Non-invasive brain stimulation technique that is used to stimulate vagal afferent projections to the nucleus of the solitary tract. Invasive VNS has been approved for the treatment of treatment-resistant depression.
  Other Names: transcutaneous auricular vagus nerve stimulation
Device: sham stimulation — Sham procedure for active transcutaneous vagus nerve stimulation
  Other Names: transcutaneous stimulation of the earlobe

SUMMARY:
Attaining goals or rewards commonly entails response costs. In light of cost and benefits, how do participants decide what effort should be put in to give it a shot? Figuratively, you may "go with your gut", but the literal contribution of the gut-brain axis in allocating effort is poorly understood to date. Here, the investigators propose to investigate non-invasive transcutaneous vagal nerve stimulation (tVNS) as a potential modulator of energy metabolism and response vigor. Since the neural mechanisms causing the diverse cognitive and behavioral effects of the stimulation remain largely elusive, the investigators will use computational modeling of instrumental behavior and determine the primary metabolic effects of the stimulation. The investigators hypothesize that tVNS will lead to activation of afferent targets in the brain. In turn, the elicited brain activation is expected to mediate the cognitive effects of the stimulation. This may affect both sides of the utility equation because anti-depressive effects may correspond to boosting the benefit of effort whereas anti-nociceptive effects may reduce perceived costs of effort. Collectively, dissecting the cognitive effects of non-invasive tVNS in healthy individuals may facilitate the more widespread use as a treatment in mental disorders that are characterized by metabolic alterations such as depression.

ELIGIBILITY:
Inclusion Criteria:

* 30 kg/m^2 > BMI > 18.5 kg/m^2

Exclusion Criteria:

lifetime

* brain injury
* coronary heart disease and occurred apoplexy
* schizophrenia
* bipolar disorder
* implants (e.g., cochlea implant)
* asthma

  12 month
* severe substance use disorders (DSM-V), except tobacco
* obessive compulsive disorder
* somatic symptom disorder
* eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Food reward ratings | during stimulation (compared to sham)
  Operationalized via visual analogue scale ratings of liking [-100 - 100] and wanting [0-100] in a food cue reactivity task
Motivation to work for rewards: frequency of button presses to gain food an monetary rewards | during stimulation (compared to sham)
  Operationalized via the relative frequency of button presses on an Xbox controller in an effort allocation task during either the first seconds of each trial (invigoration) or each complete trial (maintenance)
Reward learning: correct choices | during stimulation (compared to sham)
  Operationalized via number of correct value-based choices in a valenced go/no-go learning task
Positive and negative mood | Pre stimulation and 20 minutes post stimulation (compared to sham)
  Operationalized via visual analogue ratings (0-100) of positive and negative affect schedule mood items

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided